CLINICAL TRIAL: NCT04981158
Title: Enhanced Recovery After Lumber Laminectomy Using Combined Epidural and General Anesthesia With Tolerable Endotracheal Tube
Brief Title: Enhanced Recovery After Lumber Laminectomy Using Epidural and General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Abeer M Elnakera, MD, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZU-IRB #3225-18-12-2016
Record Dates: First submitted 2021-06-26; First posted 2021-07-28 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Recovery; Epidural Blockade; Endotracheal Tube; Laminectomy
Keywords: enhanced recovery; epidural anesthesia; tolerable endotracheal tube; general anesthesia; laminectomy
MeSH Terms: interventions — Injections, Epidural; Population Groups; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group, group I (Placebo Comparator): standard general anesthetic (GA) technique
  Interventions: Procedure: standard general anesthetic technique, control group, group I
- Epidural /GA using TET group, group II (Active Comparator): patients will undergo a single shot epidural bupivacaine (15 ml with 0.25% concentration) followed by a standard general anesthetic technique in which the trachea was intubated using tolerable endotracheal tube (TET)
  Interventions: Procedure: (Epidural /GA using tolerable endotracheal tube (TET) group, group II

INTERVENTIONS:
Procedure: (Epidural /GA using tolerable endotracheal tube (TET) group, group II — patients will undergo a single shot epidural bupivacaine (15 ml with 0.25% concentration) followed by a standard general anesthetic technique in which the trachea was intubated using TET, through its side port 2mg/kg , lidocaine 2% will be sprayed immediately after intubation when the patient is in flat supine position then the same dose of lidocaine will be repeated 10 minutes before anesthetic discontinuation.
  Arms: Epidural /GA using TET group, group II
Procedure: standard general anesthetic technique, control group, group I — patients will undergo standard general anesthesia with classic endotracheal tube
  Arms: control group, group I

SUMMARY:
Now, enhanced recovery after surgery (ERAS) is considered an essential goal to improve patient satisfaction, increase surgical workflow rate and facilitate performing different surgical procedures, including lumber laminectomy, on an ambulatory base. Different ERAS protocols have been applied and succeeded to improve recovery profile after colonic, rectal, gastric, urologic, biliary, pancreatic, and gynecologic procedures. Up to our knowledge, it is the 1st trial that will investigate the effect of combining single shot epidural blockade and general anesthesia (GA) using tolerable endotracheal tube (TET), as components for ERAS protocol for patients undergoing lumber laminectomy, on postoperative recovery profile. so the current study will be done to assess if Single shot epidural blockade and GA using TET, for patients undergoing lumber laminectomy, can enhance their postoperative recovery.

DETAILED DESCRIPTION:
The study will be carried out at anesthesia and surgical intensive care department -Zagazig University Hospitals. Patients of both sexes, assigned to a single or double level lumbar laminectomy or discectomy, will be included in the study. all patients will be preoperatively evaluated according to standard local protocol. patients, who will not be excluded, will be assigned to one of two groups: Group I (control group) patients who will undergo standard general anesthetic technique and Group II (combined general/ epidural anesthesia group (CGEA)) patients will undergo single shot epidural analgesia [by bupivacaine (15 ml with 0.25% concentration)] followed by induction of standard general anesthesia (GA) using tolerable endotracheal tube (TET)

Both groups will be compared as regard:

1. Patient recovery in the form of time to extubation, , time to achieving modified aldrete score ≥ 9 , duration of post-anesthesia care unit (PACU) stay and incidence of PACU bypass.
2. Patients' satisfaction, time to Post anesthesia discharge scoring system (PADSS) for determining home readiness ≥ 9 and incidence of hospital re-admission
3. Intra operative hemodynamic stability, blood loss, operative time and surgeon's satisfaction.
4. Postoperative pain scores and analgesic requirements.

Sample size was calculated using Epi Info 6, based on expected time to modified Aldrete score ≥ 9 in group I 13.1± 3.7 in group GA and in group II 7.9 ± 3.2 , confidence interval 95% and power of test 80%, to be 32. Eight patients will be added to compensate for dropout, so the total number of patients will be 40 patients.

All data will be collected, tabulated and statistically analyzed using SPSS 20.0 for windows (SPSS Inc., Chicago, IL, USA) and MedCalc 13 for windows (MedCalc Software bvba, Ostend, Belgium). According to the type of data qualitative data will be represented as number and percentage, parametric quantitative data will be represented by mean ± standard deviation (SD), non-parametric data will be presented as median and range and the following tests were used to test differences for significance and association of qualitative variable by Chi square test (X2). Differences between quantitative multiple by student t-test or Mann Whitney test as appropriate. P value was set at <0.05 for significant results.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) grade I-II
* body mass index (BMI) < 30 kg/m2
* assignment to a single or double level lumbar laminectomy or discectomy

Exclusion Criteria:

* Patient's refusal of the procedure
* local infection at site of catheter insertion
* recurrent disc surgery, emergency surgery
* coagulopathies
* hemoglobin <8 g/dl
* history of stroke or psychiatric disease
* baseline neurological deficit
* active upper respiratory tract infections
* history of either laryngeal / tracheal surgery or pathology
* uncontrolled hypertension or diabetes mellitus (DM), cardiac, pulmonary, hepatic or renal dysfunction
* any contraindication for study technique or medications
* being on regular steroids, opioid analgesics or alpha 2 agonists.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Time to achievement of phase I recovery criteria | the period of time (mins) starting from extubation to achievement of modified Aldrete score ≥ 9. estimated period of time 30 minutes
  time to achievement of modified Aldrete score ≥ 9 after GA or CGEA. modified aldrete score (0- 10) higher score is better score
incidence of successful PACU bypass | immediately before postoperative patient transfer out from the operating room
  number of patients who will achieve a modified Aldrete score ≥ 9 before PACU admission. modified aldrete score (0- 10) higher score is better score

SECONDARY OUTCOMES:
Time to extubation | the period of time (minutes) starting from neuromuscular reversal until endotracheal extubation. estimated period of time 15 minutes
  Time to achievement of postoperative extubation criteria (eye opening, obeying commands)
Time to achievement of phase II recovery criteria | the period of time (hours) starting from endotracheal extubation to achievement of post anesthesia discharge scoring system (PADSS) for determining home readiness ≥ 9. estimated period of time 48 hours
  Time to achievement of post anesthesia discharge scoring system (PADSS) for determining home readiness ≥ 9. PADSS (0-10). higher score is better score
incidence of persistant coughing or agitation on emergence from GA | occuring after neuromuscular reversal up to 20 mins after extubation
  persistant coughing due to tracheal irritation by endotracheal tube (ETT), agitation is defined as RSS=1
patient's rating of perioperative satisfaction | immediately before hospital discharge (after the 1st postoperative 24- 48 hrs)
  measured on a scale from 1 to 10. higher score is better score

OTHER OUTCOMES:
Time to 1st postoperative rescue analgesia | period of time (minutes) from extubation time to 1st diclofenac administration. estimated period is the 1st postoperative 6 hours
  time to 1st achievement of moderate to severe pain visual analogue score for pain (VAS)≥ 0.4. VAS for pain (0- 10). lower scores indicate better pain control
Total postoperative rescue analgesic doses required to maintain VAS for pain less than 4 | Total postoperative rescue nalbufen (mg)) requirements for 1st postoperative 24hrs
  Total postoperative rescue nalbufen (mg)) requirements
incidence of intraoperative complications | during operative period (from anesthetic induction to tracheal extubation. estimated time 2 hours
  number of patients who will suffer either intraoperative hypotension or bradycardia
incidence of postoperative complications | from extubation to home discharge. estimated time 48 hrs
  number of patients who will suffer postoperative hypotension, bradycardia, excessive sedation (RSS RSS≥ 5), new neurological deficit, postoperative nausea and vomiting (PONV) or urine retention

CONTACTS AND LOCATIONS:
Overall Officials: tarek Y Gaafar, MD, Study Chair — Zagazig University; abeer M elnakera, MD, Principal Investigator — Zagazig University; abeer H alsawy, Study Director — Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Outside US, Egypt

IPD SHARING:
Plan to Share IPD: No